CLINICAL TRIAL: NCT00512369
Title: Angiotensin, the Vascular Endothelium, and Fibrinolysis - The Effects of PAI-1 Transcriptional Regulation on Human Monocyte Function
Brief Title: Effects of PA-1 Transcriptional Regulation on Monocyte Function
Status: Terminated | Type: Observational
Why Stopped: Investigator left institution
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Douglas Vaughan, Vanderbilt University
Other Study IDs: 060286; NIH
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Atherosclerosis
Keywords: Metabolic pathways; Atherosclerosis; Monocyte Function
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Researching genetic differences in people with no prior medical conditions for better understanding of cardiac diseases through genetic research.

DETAILED DESCRIPTION:
The discovery and subsequent application of small interfering RNA (siRNA) methods to achieve individual gene silencing in mammalian cells is a robust method that is well-described and validated in mammalian cell culture systems. We will apply this technique to achieve post-transcriptional "silencing" of PAI-1 in monocytes obtained from otherwise healthy volunteers, and study the subsequent loss of this gene's function on the migratory capacity of these cells in the proposed in vitro experimental system. This concept has not yet been demonstrated in the literature, and if validated, would be a novel and fundamental description of the role of PAI-1 in human monocyte biology as related to the development of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 -50
* No current or past medical problems

Exclusion Criteria:

* Patients taking prescription drugs (hormonal birth control or herbal supplements may be taken.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese men and women
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2006-03; Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Sathyamoorthy, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States